CLINICAL TRIAL: NCT00074984
Title: Multi-Center, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Fabrazyme on Progression of Renal Disease and Significant Clinical Events in Patients With Fabry Disease
Brief Title: A Study of the Safety and Efficacy of Fabrazyme (Agalsidase Beta) as Compared to Placebo in Patients With Advanced Fabry Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Coporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGAL-008-00
Record Dates: First submitted 2003-12-24; First posted 2003-12-25 (Estimated); Results first posted 2010-12-15 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Fabry Disease
Keywords: a-Galactosidase A; aGAL; r-haGAL; Fabry; GL-3; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients randomized to placebo
  Interventions: Biological: Placebo
- Fabrazyme (agalsidase beta) (Active Comparator): Patients randomized to Fabrazyme (agalsidase beta).
  Interventions: Biological: Fabrazyme (agalsidase beta)

INTERVENTIONS:
Biological: Fabrazyme (agalsidase beta) — 1mg/kg Fabrazyme (agalsidase beta) every 2 weeks
  Other Names: Fabrazyme
  Arms: Fabrazyme (agalsidase beta)
Biological: Placebo — 1 mg/kg placebo intravenously every 2 weeks
  Arms: Placebo

SUMMARY:
People with Fabry disease have an alteration in their genetic material (DNA) which causes a deficiency of the a-galactosidase A enzyme. Fabrazyme (agalsidase beta) is a drug that helps to breakdown and remove certain types of fatty substances called "glycolipids." These glycolipids are normally present within the body in most cells. In Fabry disease, glycolipids build up in various tissues such as the liver, kidney, skin, and blood vessels because a-galactosidase A is not present, or is present in small quantities. The build up of glycolipid ("globotriaosylceramide" or "GL-3") levels in these tissues in particular is thought to cause the clinical symptoms that are common to Fabry disease. This study will test the safety and efficacy of Fabrazyme in the treatment of patients with Fabry disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients must provide written informed consent
* Patients must be at least 16 years old
* Patients must have a current diagnosis of Fabry disease and have a clinical presentation consistent of Fabry disease (decreased sweating, Fabry pain, angiokeratoma, etc.)
* Patients may not have received enzyme replacement therapy as a treatment for Fabry disease
* Patients must have a documented plasma a-galactosidase A (aGAL) activity of < 1.5 nmol/hr/mL or a documented leukocyte aGAL activity of < 4 nmol/hr/mg
* Patients must have one or more of the following: a serum creatinine measurement of 1.2 to 3 mg/dL (106.1 to 265 umol/L) OR estimated creatinine clearance < 80 mL/min only if the patient's serum creatinine measurement is < 1.2 mg/dL
* Female patients of childbearing potential must have a negative pregnancy test prior to each dosing and all female patients must use a medically accepted form of contraception

Exclusion Criteria:

* Patient has undergone or is currently scheduled for kidney transplantation or is currently on dialysis
* Patient has acute renal failure
* Patient has participated in a study employing an investigational drug within 30 days of study entry
* Patient has diabetes mellitus or presence of confounding renal disease
* Patient has a history of transient ischemic attack (TIA) or ischemic stroke within 3 months of study entry documented by mild-to-moderate neurological deficit
* Patient has critical coronary disease
* Patient has congestive heart failure
* Patient has severe residual neurological deficit that will confound the detection of new events as determined by an attending neurologist and/or Principal Investigator
* Patient is unwilling to comply with the requirements of the protocol or the patient has a medical condition, serious intercurrent illness, or extenuating circumstances that would significantly decrease study compliance, including prescribed follow-up

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2001-02; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme Coorporation
Locations (26):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of San Francisco, San Francisco, California
  - University of Connecticut Health Partners, Farmington, Connecticut
  - Oncology Hematology Association, Coral Springs, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Gene Therapy Center - Dept. of Pediatrics and Institute of Human Genetics, Minneapolis, Minnesota
  - Children's Hospital, Buffalo, New York
  - Mount Sinai School of Medicine, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Washington School of Medicine, Seattle, Washington
- Canada (3):
  - Queen Elizabeth II Health Center, Halifax, Nova Scotia
  - North York General Hospital, Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- University Hospital, Prague, Czechia
- Sopron Megyei Jogu Varos Erzsebet Korhaz, Sopron, Hungary
- Klinika Chorob Metabolicznych Instytut, Warsaw, Poland
- Hope Hospital, Manchester, United Kingdom

REFERENCES:
- [Derived] Banikazemi M, Bultas J, Waldek S, Wilcox WR, Whitley CB, McDonald M, Finkel R, Packman S, Bichet DG, Warnock DG, Desnick RJ; Fabry Disease Clinical Trial Study Group. Agalsidase-beta therapy for advanced Fabry disease: a randomized trial. Ann Intern Med. 2007 Jan 16;146(2):77-86. doi: 10.7326/0003-4819-146-2-200701160-00148. Epub 2006 Dec 18. PMID 17179052

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 252 patients were screened for entry into the study and of these, 82 patients were eligible to be enrolled.
Groups:
- Placebo: Patients randomized to placebo are administered 1 mg/kg placebo intravenously every 2 weeks.
- Fabrazyme (Agalsidase Beta): Patients randomized to Fabrazyme (agalsidase beta) are administered 1mg/kg Fabrazyme (agalsidase beta) every 2 weeks.
Period: Overall Study
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta)
Started | 31 | 51
Completed | 28 | 43
Not Completed | 3 | 8
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Patient Withdrawn Per Protocol | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta) | Total
Number analyzed (Participants) | 31 | 51 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 49 | 80
  >=65 years | 0 | 2 | 2
Age, Customized [Number; unit: participants]
  <40 years | 8 | 11 | 19
  ≥40 years | 23 | 40 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (9.23) | 46.9 (9.75) | 45.9 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 27 | 45 | 72
Race/Ethnicity [Number; unit: participants]
  Caucasian | 27 | 45 | 72
  Black | 0 | 1 | 1
  Hispanic | 2 | 3 | 5
  Asian | 1 | 1 | 2
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing a Clinically Significant Renal, Cardiac or Cerebrovascular Event and/or Death in Fabrazyme (Agalsidase Beta) Patients as Compared to Placebo Patients
Description: The primary efficacy endpoint was the time to the first occurrence of a clinically significant renal (33% increase in serum creatinine, dialysis or transplant), cardiac (myocardial infarction, significant change in cardiac status, i.e., angina, congestive heart failure or symptomatic arrhythmia requiring medication or surgery) or cerebrovascular (stroke or transient ischemic attack) event and/or death (due to any cause) in Fabrazyme (agalsidase beta) patients as compared to placebo patients.
Time Frame: up to 35 months
Population: The Intent-to-treat (ITT) population consists of all 82 patients who were randomized, enrolled, and received at least one infusion of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta)
Number analyzed (Participants) | 31 | 51
participants
  Participants with a clinical event | 13 | 14
  Participants with no clinical event | 18 | 37
Statistical Analysis 1: Comparison: Placebo vs Fabrazyme (Agalsidase Beta); Test type: Superiority or Other; p = 0.1449, Log Rank; Comparison is based on a 2-sided log-rank test; Hazard Ratio (HR) = 0.574, 95% CI 2-sided [0.269 to 1.222]
Statistical Analysis 2: Comparison: Placebo vs Fabrazyme (Agalsidase Beta); Time to First Primary Endpoint Adjusting for Baseline Proteinuria using Cox Proportional Hazards Model; Test type: Superiority or Other; p = 0.0577, Wald Test; Cox Proportional Hazard = 0.465, 95% CI 2-sided [0.211 to 1.025]

2. Secondary Outcome: Number of Participants Experiencing a Renal Event in Fabrazyme (Agalsidase Beta) Patients as Compared to Placebo Patients
Description: Time to a clinically significant renal event (33% increase in serum creatinine, dialysis or transplant) in Fabrazyme (agalsidase beta) patients as compared to placebo patients.
Time Frame: up to 35 months
Population: The Intent-to-treat population consisted of all 82 patients who were randomized, enrolled, and received at least one infusion of study medication.
Measure: Number; unit: participants
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta)
Number analyzed (Participants) | 31 | 51
participants
  Participants with a Renal event | 7 | 10
  Participants with no Renal event | 24 | 41
Statistical Analysis 1: Comparison: Placebo vs Fabrazyme (Agalsidase Beta); Analysis of Time to First Renal Event for ITT population; Test type: Superiority or Other; p = 0.5261, Log Rank; 2-sided log-rank test; Hazard Ratio (HR) = 0.732, 95% CI 2-sided [0.278 to 1.927]

3. Secondary Outcome: Slope of Estimated Glomerular Filtration Rate (eGFR) Comparing Placebo vs Fabrazyme (Agalsidase Beta) Patients
Description: Summary of slopes of eGFR by baseline eGFR subgroups (>60 and <=60 mL/min/1.73m^2/year) comparing Placebo vs Fabrazyme (agalsidase beta) Patients.
Time Frame: up to 35 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2/year
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta)
Number analyzed (Participants) | 31 | 51
mL/min/1.73m^2/year
  eGFR Total | -3.62 (3.38) | -3.25 (2.92)
  Baseline eGFR >60 | -5.09 (3.52) | -1.51 (2.85)
  Baseline eGFR <= 60 | -3.02 (3.21) | -4.20 (2.52)

4. Secondary Outcome: Slope of Inverse Serum Creatinine Values Comparing Placebo vs Fabrazyme (Agalsidase Beta)Patients
Description: Summary of slopes of inverse serum creatinine by baseline serum creatinine subgroups (> or <= 1.5 mg/dL) comparing Placebo vs Fabrazyme (agalsidase beta) patients.
Time Frame: up to 35 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: dL/mg/year
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta)
Number analyzed (Participants) | 31 | 51
dL/mg/year
  Total | -0.038 (0.037) | -0.036 (0.035)
  Baseline Serum Creatinine > 1.5 | -0.043 (0.030) | -0.050 (0.028)
  Baseline Serum Creatinine <= 1.5 | -0.033 (0.043) | -0.022 (0.035)

5. Secondary Outcome: Neuropathic Pain as Assessed by Question 12 of the Brief Pain Inventory (BPI) Questionnaire (Pain at Its Worst)
Description: Neuropathic pain was assessed by Question 12 of the Brief Pain Inventory (BPI) Questionnaire on a scale of 0 (no pain) to 10 (pain as bad as you can imagine)
Time Frame: at 24 months
Population: Intent-to-treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Fabrazyme (Agalsidase Beta)
Number analyzed (Participants) | 31 | 51
units on a scale
  Baseline (n=30, n=48) | 2.2 (3.0) | 2.7 (3.1)
  2 years (n=7, n=18) | 4.4 (3.6) | 2.7 (3.2)
  Change from baseline to 2 years (n=7, n=17) | 0.9 (3.0) | -0.8 (3.2)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Groups:
- Fabrazyme (Agalsidase Beta): Patients randomized to Fabrazyme(agalsidase beta) are administered 1mg/kg Fabrazyme (agalsidase beta) every 2 weeks.
- Total: All patients.
Arm/Group | Fabrazyme (Agalsidase Beta) | Placebo | Total
Serious Adverse Events (participants affected / at risk) | 18/51 | 12/31 | 30/82
Other Adverse Events (participants affected / at risk) | 51/51 | 29/31 | 80/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme (Agalsidase Beta) (N=51) | Placebo (N=31) | Total (N=82)
Angina pectoris (Cardiac disorders) | 0 | 1 | 1
Angina unstable (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3
Atrioventricular block second degree (Cardiac disorders) | 1 | 1 | 2
Bradycardia (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 2
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Chest pain (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 2 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1
Streptococcal infection (Infections and infestations) | 1 | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Medical device complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural hypertension (Injury, poisoning and procedural complications) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 1
Skin test positive (Investigations) | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1
Affective disorder (Psychiatric disorders) | 0 | 1 | 1
Alcoholism (Psychiatric disorders) | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Nephritis interstitial (Renal and urinary disorders) | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Drug therapy changed (Surgical and medical procedures) | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme (Agalsidase Beta) (N=51) | Placebo (N=31) | Total (N=82)
Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 8
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1
Aortic valve sclerosis (Cardiac disorders) | 0 | 2 | 2
Arrhythmia (Cardiac disorders) | 2 | 0 | 2
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 2 | 3
Bradycardia (Cardiac disorders) | 3 | 2 | 5
Bundle branch block (Cardiac disorders) | 0 | 1 | 1
Bundle branch block right (Cardiac disorders) | 3 | 0 | 3
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1
Dilatation atrial (Cardiac disorders) | 2 | 3 | 5
Heart valve insufficiency (Cardiac disorders) | 1 | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 1 | 2
Mitral valve prolapse (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Palpitations (Cardiac disorders) | 4 | 1 | 5
Sinus arrhythmia (Cardiac disorders) | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 2
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0 | 2
Tachyarrhythmia (Cardiac disorders) | 1 | 0 | 1
Tachycardia (Cardiac disorders) | 3 | 1 | 4
Ventricular dysfunction (Cardiac disorders) | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 2 | 3
Ventricular hypertrophy (Cardiac disorders) | 2 | 3 | 5
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 2
Ventricular wall thickening (Cardiac disorders) | 2 | 0 | 2
Cerumen impaction (Ear and labyrinth disorders) | 1 | 0 | 1
Deafness (Ear and labyrinth disorders) | 1 | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 1
Ear canal erythema (Ear and labyrinth disorders) | 0 | 1 | 1
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 2 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 2 | 2 | 4
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 1
Hypoacusis (Ear and labyrinth disorders) | 3 | 0 | 3
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1 | 1
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 6 | 1 | 7
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 3
Hyperparathyroidism (Endocrine disorders) | 1 | 0 | 1
Hypothalamo-pituitary disorders (Endocrine disorders) | 0 | 1 | 1
Binocular eye movement disorder (Eye disorders) | 2 | 0 | 2
Blepharitis (Eye disorders) | 1 | 0 | 1
Blepharospasm (Eye disorders) | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 1
Cataract subcapsular (Eye disorders) | 0 | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 1
Eye irritation (Eye disorders) | 1 | 0 | 1
Eye pain (Eye disorders) | 2 | 0 | 2
Eyelid oedema (Eye disorders) | 1 | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0 | 1
Retinopathy (Eye disorders) | 1 | 0 | 1
Scleral haemorrhage (Eye disorders) | 1 | 0 | 1
Vision blurred (Eye disorders) | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 8 | 4 | 12
Abdominal pain lower (Gastrointestinal disorders) | 3 | 0 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 7
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 1 | 4
Defaecation urgency (Gastrointestinal disorders) | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 12 | 7 | 19
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 5
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 1
Faeces pale (Gastrointestinal disorders) | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 3 | 1 | 4
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal hypermotility (Gastrointestinal disorders) | 1 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 1
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 2 | 0 | 2
Lip blister (Gastrointestinal disorders) | 0 | 1 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 9 | 10 | 19
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1
Stomach discomfort (Gastrointestinal disorders) | 4 | 0 | 4
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1
Tooth disorder (Gastrointestinal disorders) | 0 | 1 | 1
Toothache (Gastrointestinal disorders) | 4 | 2 | 6
Uvulitis (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 14 | 10 | 24
Adverse event (General disorders) | 8 | 3 | 11
Asthenia (General disorders) | 5 | 2 | 7
Axillary pain (General disorders) | 1 | 0 | 1
Catheter site haematoma (General disorders) | 1 | 0 | 1
Catheter site pain (General disorders) | 0 | 1 | 1
Catheter site related reaction (General disorders) | 1 | 0 | 1
Chest discomfort (General disorders) | 3 | 1 | 4
Chest pain (General disorders) | 5 | 5 | 10
Chills (General disorders) | 20 | 6 | 26
Cyst (General disorders) | 0 | 1 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1 | 1
Face oedema (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 17 | 4 | 21
Feeling cold (General disorders) | 4 | 1 | 5
Feeling hot (General disorders) | 2 | 1 | 3
Feeling hot and cold (General disorders) | 1 | 0 | 1
Feeling jittery (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 1 | 0 | 1
Influenza like illness (General disorders) | 3 | 1 | 4
Infusion site reaction (General disorders) | 2 | 2 | 4
Injection site thrombosis (General disorders) | 1 | 0 | 1
Irritability (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 2 | 1 | 3
Oedema peripheral (General disorders) | 12 | 9 | 21
Pain (General disorders) | 12 | 7 | 19
Pitting oedema (General disorders) | 2 | 0 | 2
Pyrexia (General disorders) | 18 | 9 | 27
Suprapubic pain (General disorders) | 1 | 0 | 1
Thirst (General disorders) | 1 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 2 | 0 | 2
Multiple allergies (Immune system disorders) | 0 | 1 | 1
Bronchitis (Infections and infestations) | 3 | 2 | 5
Bronchitis acute (Infections and infestations) | 1 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Conjunctivitis infective (Infections and infestations) | 1 | 0 | 1
Dental caries (Infections and infestations) | 0 | 1 | 1
Ear infection (Infections and infestations) | 1 | 2 | 3
Fungal infection (Infections and infestations) | 4 | 0 | 4
Gastroenteritis (Infections and infestations) | 3 | 2 | 5
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1
Gingival abscess (Infections and infestations) | 0 | 1 | 1
Gingival infection (Infections and infestations) | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 2 | 2
Influenza (Infections and infestations) | 6 | 4 | 10
Kidney infection (Infections and infestations) | 1 | 0 | 1
Labyrinthitis (Infections and infestations) | 0 | 1 | 1
Localised infection (Infections and infestations) | 2 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 9 | 1 | 10
Mastoiditis (Infections and infestations) | 1 | 1 | 2
Nail tinea (Infections and infestations) | 1 | 0 | 1
Nasopharyngitis (Infections and infestations) | 17 | 6 | 23
Oral candidiasis (Infections and infestations) | 0 | 1 | 1
Otitis externa fungal (Infections and infestations) | 0 | 1 | 1
Otitis media (Infections and infestations) | 1 | 1 | 2
Pharyngitis (Infections and infestations) | 1 | 1 | 2
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 1
Postoperative infection (Infections and infestations) | 2 | 0 | 2
Prostate infection (Infections and infestations) | 1 | 0 | 1
Rectal abscess (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 2
Sinusitis (Infections and infestations) | 6 | 3 | 9
Skin infection (Infections and infestations) | 0 | 1 | 1
Tooth abscess (Infections and infestations) | 4 | 1 | 5
Upper respiratory tract infection (Infections and infestations) | 16 | 8 | 24
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 3
Vaginal candidiasis (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 5 | 0 | 5
Viral upper respiratory tract infection (Infections and infestations) | 6 | 0 | 6
Animal scratch (Injury, poisoning and procedural complications) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 2 | 1 | 3
Back injury (Injury, poisoning and procedural complications) | 3 | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 4 | 2 | 6
Ear canal abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 1
Electric shock (Injury, poisoning and procedural complications) | 1 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 7 | 1 | 8
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 4
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 2
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 2
Open wound (Injury, poisoning and procedural complications) | 1 | 0 | 1
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Post procedural nausea (Injury, poisoning and procedural complications) | 1 | 0 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 6 | 0 | 6
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 2 | 1 | 3
Thermal burn (Injury, poisoning and procedural complications) | 2 | 0 | 2
Tooth fracture (Injury, poisoning and procedural complications) | 3 | 1 | 4
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Albumin urine present (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 2 | 0 | 2
Blood bicarbonate decreased (Investigations) | 7 | 4 | 11
Blood bilirubin increased (Investigations) | 1 | 0 | 1
Blood calcium decreased (Investigations) | 3 | 1 | 4
Blood chloride increased (Investigations) | 2 | 0 | 2
Blood creatinine increased (Investigations) | 6 | 2 | 8
Blood glucose increased (Investigations) | 0 | 1 | 1
Blood phosphorus increased (Investigations) | 1 | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 1
Blood potassium increased (Investigations) | 1 | 2 | 3
Blood pressure decreased (Investigations) | 1 | 2 | 3
Blood pressure increased (Investigations) | 6 | 2 | 8
Blood sodium decreased (Investigations) | 1 | 1 | 2
Blood triglycerides increased (Investigations) | 1 | 0 | 1
Blood urea increased (Investigations) | 3 | 1 | 4
Blood uric acid increased (Investigations) | 2 | 1 | 3
Body temperature increased (Investigations) | 1 | 1 | 2
Cardiac murmur (Investigations) | 2 | 1 | 3
Cardiac stress test abnormal (Investigations) | 1 | 2 | 3
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 1
Echocardiogram abnormal (Investigations) | 0 | 1 | 1
Ejection fraction decreased (Investigations) | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 1 | 1
Electrocardiogram ST segment abnormal (Investigations) | 3 | 2 | 5
Electrocardiogram ST segment depression (Investigations) | 1 | 0 | 1
Electrocardiogram ST-T segment abnormal (Investigations) | 1 | 0 | 1
Electrocardiogram T wave amplitude increased (Investigations) | 0 | 1 | 1
Electrocardiogram T wave inversion (Investigations) | 2 | 0 | 2
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 1
Haematocrit decreased (Investigations) | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 0 | 3
Heart rate decreased (Investigations) | 1 | 0 | 1
Heart rate increased (Investigations) | 2 | 1 | 3
Heart rate irregular (Investigations) | 1 | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1
Nuclear magnetic resonance imaging abnormal (Investigations) | 1 | 0 | 1
Occult blood positive (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 1
Platelet count increased (Investigations) | 1 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 1
Prothrombin time ratio increased (Investigations) | 1 | 0 | 1
Red blood cell count decreased (Investigations) | 2 | 0 | 2
Red blood cells urine positive (Investigations) | 3 | 2 | 5
Right ventricular systolic pressure increased (Investigations) | 1 | 0 | 1
Tandem gait test abnormal (Investigations) | 0 | 2 | 2
Vibration test abnormal (Investigations) | 0 | 1 | 1
Weight decreased (Investigations) | 1 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 2 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 3
Gout (Metabolism and nutrition disorders) | 3 | 2 | 5
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 2 | 3
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 14
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 4 | 19
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 2 | 8
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1 | 8
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 5 | 18
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Epithelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 1
Burning sensation (Nervous system disorders) | 2 | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 2 | 4
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 1
Coordination abnormal (Nervous system disorders) | 2 | 0 | 2
Dizziness (Nervous system disorders) | 13 | 4 | 17
Dysgeusia (Nervous system disorders) | 1 | 0 | 1
Encephalomalacia (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 21 | 8 | 29
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 8 | 4 | 12
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 2 | 2
Mental impairment (Nervous system disorders) | 0 | 1 | 1
Muscle contractions involuntary (Nervous system disorders) | 0 | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 2
Nystagmus (Nervous system disorders) | 0 | 1 | 1
Paraesthesia (Nervous system disorders) | 18 | 8 | 26
Reflexes abnormal (Nervous system disorders) | 0 | 1 | 1
Sciatica (Nervous system disorders) | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Syncope vasovagal (Nervous system disorders) | 1 | 0 | 1
Tremor (Nervous system disorders) | 2 | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 4 | 3 | 7
Depressed mood (Psychiatric disorders) | 2 | 0 | 2
Depression (Psychiatric disorders) | 4 | 0 | 4
Flat affect (Psychiatric disorders) | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 6 | 2 | 8
Mood altered (Psychiatric disorders) | 1 | 0 | 1
Panic attack (Psychiatric disorders) | 1 | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 0 | 3 | 3
Azotaemia (Renal and urinary disorders) | 1 | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 0 | 2
Haematuria (Renal and urinary disorders) | 0 | 3 | 3
Micturition disorder (Renal and urinary disorders) | 1 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 5 | 0 | 5
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0 | 1
Urethral stricture (Renal and urinary disorders) | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 1
Breast discharge (Reproductive system and breast disorders) | 1 | 0 | 1
Breast discomfort (Reproductive system and breast disorders) | 1 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 1
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 1
Scrotal angiokeratoma (Reproductive system and breast disorders) | 1 | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 1
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 11 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 5
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 7 | 20
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 18
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 10
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 9
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Angiokeratoma (Skin and subcutaneous tissue disorders) | 3 | 2 | 5
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Anhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 1 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 4
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2 | 6
Pruritus allergic (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 4 | 11
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 1 | 3
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Flushing (Vascular disorders) | 2 | 1 | 3
Hot flush (Vascular disorders) | 3 | 1 | 4
Hypertension (Vascular disorders) | 2 | 3 | 5
Hypotension (Vascular disorders) | 2 | 3 | 5
Lymphoedema (Vascular disorders) | 1 | 0 | 1
Pallor (Vascular disorders) | 1 | 1 | 2
Peripheral coldness (Vascular disorders) | 2 | 1 | 3
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 1
Steal syndrome (Vascular disorders) | 1 | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.